CLINICAL TRIAL: NCT04579913
Title: A Multi-center, International Prospective Follow up Study to Assess the Safety and Efficacy of the iTind Procedure After Three to Five Years of Follow Up
Brief Title: A Multi-center, International Prospective Follow up Study
Status: Terminated | Type: Observational
Why Stopped: Covid-19
Sponsor: Medi-Tate Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MT-03A
Record Dates: First submitted 2020-09-29; First posted 2020-10-08 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- iTind subjects: Patient who participated previously in the MT-03 study in the iTind arm
  Interventions: Other: Review of medical history, administration of questionnaires, uroflowmetry and PVR as measured by ultrasound

INTERVENTIONS:
Other: Review of medical history, administration of questionnaires, uroflowmetry and PVR as measured by ultrasound — Administration of questionnaires to assess patient LUTS, quality of life, sexual behavior and erectile function, in addition to performing PVR and uroflow tests.

SUMMARY:
The study objective is to assess the safety and efficacy of iTind three to five years following treatment.

DETAILED DESCRIPTION:
This study will recruit patients who participated in the MT-03 study in the iTind arm to assess the safety and efficacy of the iTind procedure at three to five years following treatment as demonstrated by reduction of symptoms measured by IPSS and QoL and improvement of functional parameters as measured by peak urinary flow and PVR. Sexual and erectile function will also be assessed alongside the incidence of any related late occurring adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Subject signed informed consent form (ICF)
2. Subject who had participated in the MT-03 study in the iTind arm
3. Subject able to comply with the study protocol.

Exclusion Criteria:

1. Any anatomical or physiological condition that in the opinion of the investigator likely to impede successful completion of the study
2. Patients that are known to have had undergone an alternative surgical procedure for BPH during MT-03 study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient who participated in the MT-03 study in the iTind arm who had not undergone an alternative procedure for BPH during the first 12 month follow-up period and who is willing to participate in the current follow up study.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
iTind Durability | 36 months post procedure
  The primary endpoint of the study is time to first alternative surgical BPH intervention, defined as the time (in months) from the iTind procedure to intervention.
iTind Durability | 48 months post procedure
  The primary endpoint of the study is time to first alternative surgical BPH intervention, defined as the time (in months) from the iTind procedure to intervention.
iTind Durability | 60 months post procedure
  The primary endpoint of the study is time to first alternative surgical BPH intervention, defined as the time (in months) from the iTind procedure to intervention.

SECONDARY OUTCOMES:
iTind Efficacy | 36 months post procedure
  Change from baseline in IPSS
iTind Efficacy | 48 months post procedure
  Change from baseline in IPSS
iTind Efficacy | 60 months post procedure
  Change from baseline in IPSS
iTind Efficacy | 36 months post procedure
  Change from baseline in Qmax
iTind Efficacy | 48 months post procedure
  Change from baseline in Qmax
iTind Efficacy | 60 months post procedure
  Change from baseline in Qmax
iTind Safety | 36 months post procedure
  Safety will be assessed by the rate of complications attributed to iTind since the last recorded follow up from MT-03 study
iTind Safety | 48 months post procedure
  Safety will be assessed by the rate of complications attributed to iTind since the last recorded follow up from MT-03 study
iTind Safety | 60 months post procedure
  Safety will be assessed by the rate of complications attributed to iTind since the last recorded follow up from MT-03 study

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Manhattan Medical research, Manhattan, New York
  - Premier Urology Group, New York, New York
  - Lenox Hill Hospital, New York, New York
- Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company website — https://www.itind.com/